CLINICAL TRIAL: NCT06732518
Title: Clinical Study to Evaluate the Anti-cavity Efficacy of Three Dentifrices Using an Intra-oral Enamel Demineralization - Remineralization In-Situ Model
Brief Title: Evaluation of the Anti-cavity Efficacy of Three Dentifrices Using an Intra-oral Enamel Demineralization - Remineralization In-Situ Model
Acronym: REPAIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Collaborators: Federal University of Alagoas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CRO-2024-04-DEM-REM-BZ-BG
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-04

CONDITIONS: Enamel Lesions; Demineralization, Tooth; Remineralization; Dental Cavity
Keywords: enamel demineralization-remineralization; fluoride toothpaste; enamel microhardness
MeSH Terms: conditions — Tooth Demineralization; Dental Caries

STUDY DESIGN:
Intervention Model Description: This is a Phase III, randomized, one-center, crossover group, triple blind, clinical study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this clinical trial, masking involves several key roles to ensure unbiased results. The Participant, Care Provider, Investigator, and Outcomes Assessor are all masked in this triple-blind study. This means that the participants do not know which group they have been assigned to, the care providers administering the treatments are unaware of the specific products being used by each participant, the investigators conducting the study do not know the group assignments, and the outcomes assessors evaluating the results are blind to the treatment allocations. This comprehensive masking approach is designed to minimize any potential biases and maintain the integrity of the study results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fluoride toothpaste (Experimental): Subjects will brush using a fluoride toothpaste containing 1000 ppm MFP and 1.5% arginine in a PCC/RNCC base and a soft bristle toothbrush
  Interventions: Drug: Fluoride Toothpaste; Device: Toothbrush
- Fluoride free toothpaste in a chalk base (Active Comparator): Subjects will brush using a fluoride free toothpaste in a chalk base with herbal ingredients and a soft bristle toothbrush
  Interventions: Drug: Fluoride free toothpaste in a chalk base; Device: Toothbrush
- Fluoride free toothpaste in a PCC/RNCC base (Active Comparator): This is a negative control group in which subjects will brush using a fluoride free toothpaste in a PCC/RNCC base and a soft bristle toothbrush
  Interventions: Drug: Fluoride free toothpaste in a PCC/RNCC base; Device: Toothbrush
- Washout (Other): This is a washout group in which subjects will brush using a fluoride free toothpaste in a PCC/RNCC base and a soft bristle toothbrush for 9 days, between the treatment phases
  Interventions: Drug: Fluoride free toothpaste in a PCC/RNCC base; Device: Toothbrush

INTERVENTIONS:
Drug: Fluoride Toothpaste — Fluoride toothpaste containing 1000 ppm MFP and 1.5% arginine in a PCC/RNCC base
  Arms: Fluoride toothpaste
Drug: Fluoride free toothpaste in a chalk base — Fluoride free toothpaste in a chalk base with herbal ingredients
  Arms: Fluoride free toothpaste in a chalk base
Drug: Fluoride free toothpaste in a PCC/RNCC base — Fluoride free toothpaste in a PCC/RNCC base
  Arms: Fluoride free toothpaste in a PCC/RNCC base; Washout
Device: Toothbrush — A commercially available adult soft bristle toothbrush

SUMMARY:
Clinical study to evaluate the anti-cavity efficacy of three dentifrices using an intra-oral enamel Demineralization - Remineralization In-Situ Model. This is a Phase III, single-center, triple-blind with a crossover design. It involves 36 participants aged between 18 and 70, randomized into 3 different groups + a washout group, and spans 6 weeks.

DETAILED DESCRIPTION:
This clinical study aims to evaluate the anti-cavity efficacy of dentifrices using an intra-oral enamel demineralization-remineralization in-situ model. It is a Phase III, randomized, triple-blind, crossover study involving 36 participants aged 18 to 70. Participants will use an intra-oral appliance with a steel mesh holding bovine enamel blocks, properly disinfected before using. Participants will be divided into three groups of treatment: one using a fluoride-free toothpaste with a chalk base and herbal ingredients, another using a fluoride toothpaste containing 1000 ppm MFP and 1.5% arginine in a PCC/RNCC base, and a negative control group using a fluoride-free toothpaste in a PCC/RNCC base. Each participant will receive a soft-bristle toothbrush and will be instructed to brush twice daily for 6 weeks. Additionally, between the treatment phases (5 days), 9-day washout phases will occur, during which participants will use a fluoride-free toothpaste in a PCC/RNCC base. Subjects will undergo baseline visit, visit 2 - washout I (9 days), visit 3 - treatment phase I (5 days), visit 4- washout II, visit 5- treatment phase II, visit 6 - washout III, visit 7 - treatment phase III, visit 8 - final visit. The primary outcome will be enamel microhardness, measured before and after treatment, to assess changes in microhardness. The expected outcome is the confirmation of the alternative hypothesis, which predicts a reduction in the percentage of mineral loss from the surface of bovine enamel after using dentifrices containing 1000 ppm MFP with 1.5% arginine or herbal ingredients for five days each, compared to the control group. The percentage of mineral loss on the tooth surface relative to baseline will be used to quantify the extent of reduction in enamel demineralization. A two factor ANCOVA using the baseline as the covariate will be conducted to determine if a significant treatment effect exists. Adverse events and compliance will be closely monitored, with strict confidentiality maintained for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, between 18-70 years of age (inclusive);
* Informed Consent Form signed and availability for the duration of the study;
* Good general health (absence of any condition that, in the opinion of the Principal Investigator, might constitute a risk to the subject while participating in the study. Examples include heart problems, valve/hip replacements, etc);
* Willingness to provide information related to their medical history;
* Minimum of 20 uncrowned permanent natural teeth (excluding third molars); Normal salivary flow;
* Willingness to wear an intra-oral appliance all day as instructed except when eating and drinking.

Exclusion Criteria:

* Oral pathology, chronic disease, or a history of allergy to testing products;
* Subject using anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory medication or daily analgesics within one month prior to the start of the study or scheduled to start such intake during the course of the study;
* Subject participating in any other clinical study;
* Subject pregnant or breastfeeding;
* Subject allergic to oral care products, personal care consumer products, or their ingredients;
* Extended use of antibiotics or therapeutic mouthwash any time during the three months prior to entry into the study;
* A medical history reporting that the subject has a current systemic or autoimmune disease, such as diabetes, lupus, etc.;
* Ongoing use of medications known to affect the gingival tissues (i.e. calcium channel blockers, phenytoin, cyclosporine);
* Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone). Pocket depth equal or greater than 4 mm
* Five or more decayed, untreated dental sites (cavities);
* Current smokers and subjects with a history of alcohol or drug abuse;
* Dental work prevents wearing of the appliance or a reported need to wear a night guard.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Microhardness change | 6 weeks
  The primary measured response will be a change in indentation length in the intra-oral appliance before and after treatment for microhardness. The indentation length will be used to calculate a hardness value. The percentage of mineral loss on the bovine tooth enamel surface relative to baseline will be used to quantify the extent of reduction in enamel demineralization.

CONTACTS AND LOCATIONS:
Overall Officials: Natanael Silva, PhD, Principal Investigator — Federal University of Alagoas
Locations (1):
- Federal University of Alagoas, Maceió, Alagoas, Brazil

IPD SHARING:
Plan to Share IPD: No